CLINICAL TRIAL: NCT06308887
Title: Comparison of the Effectiveness of Ultrasound-Guided Perimeniscal Steroid and Dextrose Injections in Knee Osteoarthritis
Brief Title: Comparison of Ultrasound-Guided Perimeniscal Steroid and 5% Dextrose Injections in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Gamze Gul Gulec, Doctor, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Gonarthrosis; Meniscus; Degeneration; Pain, Chronic
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — triamcinolone hexacetonide; Triamcinolone; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): patients who had perimeniscal 5 % dextrose injection
  Interventions: Drug: Dextrose 5% in water
- Group 2 (Active Comparator): patients who had perimeniscal triamcinolone injection
  Interventions: Drug: Triamcinolone Hexacetonide

INTERVENTIONS:
Drug: Triamcinolone Hexacetonide — Ultrasound-guided periarticular (perimeniscal) injection: The injections were administered using ultrasonic guidance on the longitudinal axis while the patient was in a supine position with the knee flexed at approximately 20°-30°. The transducer was positioned longitudinally in the region where extrusion was seen along the medial collateral ligament. Subsequently, employing a free-hand method, a 0.60x60 mm 23 G needle was inserted directly into the meniscus wall with the use of sonographic guidance. After the needle made contact with the medial meniscus wall, it was pulled back by 1 mm and placed between the medial collateral ligament and the medial meniscus, and a dose of 0.5 mg/5 ml of triamcinolone acetonide was injected.
  Other Names: kenacort
  Arms: Group 2
Drug: Dextrose 5% in water — Ultrasound-guided periarticular (perimeniscal) injection: The injections were administered using ultrasonic guidance on the longitudinal axis while the patient was in a supine position with the knee flexed at approximately 20°-30°. The transducer was positioned longitudinally in the region where extrusion was seen along the medial collateral ligament. Subsequently, employing a free-hand method, a 0.60x60 mm 23 G needle was inserted directly into the meniscus wall with the use of sonographic guidance. After the needle made contact with the medial meniscus wall, it was pulled back by 1 mm and placed between the medial collateral ligament and the medial meniscus, and a dose of 5 ml of 5% dextrose was injected.
  Arms: Group 1

SUMMARY:
Introduction: The primary goal of treating knee osteoarthritis is to reduce pain and improve the patient's quality of life. Medial meniscal extrusion is a condition that is linked to pain and disability in knee osteoarthritis and can be identified through ultrasound. For patients with medial meniscal extrusion, perimeniscal corticosteroid injection has been shown to be a helpful addition to primary treatment for moderate to severe pain relief. Dextrose prolotherapy has also been found to provide periarticular benefits for knee osteoarthritis. This study aims to compare the effectiveness of ultrasound-guided perimeniscal corticosteroid and perimeniscal dextrose injections in patients with osteoarthritis, medial knee pain, and medial meniscal extrusion.

Method: Patients with medial knee pain and meniscal extrusion were randomly divided into two groups using the double-block randomization method. Group 1 included 15 patients who were administered an ultrasound-guided perimeniscal steroid injection, while Group 2 included 16 patients who were administered an ultrasound-guided perimeniscal dextrose injection. The patients' pain levels were evaluated using the Visual Analog Pain Scale (VAS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) before and one week, one month, and three months after the injection.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2-4 knee osteoarthritis,
* Aged 40 to 79
* Chronic medial knee pain persisting for more than 3 months.
* Ultrasound screening found medial meniscal extrusion of more than 3 mm
* A Visual Analog Scale (VAS) score of at least 4.

Exclusion Criteria:

a skin infection at the injection site, a prior history of inflammatory arthropathy, a prior history of knee injection within the last 3 months, knee synovitis pes anserine bursitis scheduled for surgery

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | At the beginning, 1.,4., 12. week
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression or compare pain severity between patients with similar conditions.VAS is comprised of a horizontal line of 10 cm in length. A measurement of 0 cm indicates the absence of pain, whereas a measurement of 10 cm signifies the most severe pain that one can conceive. Patients are instructed to assess the intensity of discomfort by indicating a point on this line.

SECONDARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index | At the beginning, 1.,4., 12. week
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of hip and knee osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain, stiffness, and physical function. The test questions are scored on a scale of 0-4, which corresponds to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function. Usually, a sum of the scores for all three subscales gives a total WOMAC score, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Özmen, MD, Study Chair — İstanbul Physical Medicine and Rehabilitation Hospital
Locations (1):
- Gamze Gül Güleç, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Sante L, Venditto T, Ioppolo F, Paoloni M, Mangone M, Alviti F. Ultrasound guided injection of a painful knee osteoarthritis with medial meniscus extrusion: a case series study. Muscles Ligaments Tendons J. 2017 Sep 18;7(2):331-337. doi: 10.11138/mltj/2017.7.2.331. eCollection 2017 Apr-Jun. PMID 29264345
- [Background] Bayat M, Hojjati F, Boland Nazar NS, Modabberi M, Rahimi MS. Comparison of Dextrose Prolotherapy and Triamcinolone Intraarticular Injection on Pain and Function in Patients with Knee Osteoarthritis - A Randomized Clinical Trial. Anesth Pain Med. 2023 Apr 8;13(2):e134415. doi: 10.5812/aapm-134415. eCollection 2023 Apr. PMID 37601963
- [Background] Robinson RL, Schnitzer TJ, Barlow S, Berry M, Bushmakin AG, Cappelleri JC, Tive L, Jackson J, Jackson J, Viktrup L. Satisfaction with Medications Prescribed for Osteoarthritis: A Cross-Sectional Survey of Patients and Their Physicians in the United States. Pain Ther. 2022 Mar;11(1):191-208. doi: 10.1007/s40122-021-00350-0. Epub 2022 Jan 13. PMID 35028917
- [Background] Finan PH, Buenaver LF, Bounds SC, Hussain S, Park RJ, Haque UJ, Campbell CM, Haythornthwaite JA, Edwards RR, Smith MT. Discordance between pain and radiographic severity in knee osteoarthritis: findings from quantitative sensory testing of central sensitization. Arthritis Rheum. 2013 Feb;65(2):363-72. doi: 10.1002/art.34646. PMID 22961435